CLINICAL TRIAL: NCT06817564
Title: Effects of an AI-driven Personalized Exercise Feedback Program on Exercise Adherence and Health Outcomes in Patients with Traumatic Brain Injury
Brief Title: AI-driven Personalized Exercise Feedback Program on Exercise Adherence in Traumatic Brain Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Hui-Hsun Chiang, Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AI feedback digital exercise
Record Dates: First submitted 2025-01-20; First posted 2025-02-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury; Exercise; AI (Artificial Intelligence); Digital Health
Keywords: AI-Driven Personalized Exercise Program
MeSH Terms: conditions — Brain Injuries, Traumatic; Motor Activity

STUDY DESIGN:
Intervention Model Description: Phase 2: Evaluate the feasibility, acceptability, and preliminary effectiveness of the AI-PEF in improving patient outcomes.
  Phase 3: Examine the impact of the AI-PEF on exercise adherence and health outcomes
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Physicians are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AI-PEF (Experimental): the AI-PEF group, receiving a machine learning-powered personalized exercise program.
  Interventions: Behavioral: AI-PEF
- Theory-based digital exercise (Experimental): Theory-based digital exercise group, engaging in structured digital exercise without machine learning- powered feedback.
  Interventions: Behavioral: Theory-based digital exercise
- Active control group (Active Comparator): the Active control group, receiving general exercise recommendations as part of standard care in a 1:1:1 ratio.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: AI-PEF — Participants will follow a 12-week walking program with five 30-minute sessions per week, progressively increasing intensity based on heart rate and effort indices. Garmin fitness trackers will monitor adherence and intensity. Remote guidance will support participants via weekly digital health messages on the LINE app, offering personalized feedback, goal reinforcement, and lifestyle recommendations. Participants will also receiThese AI feedback implementations will be tailored to complement the in-person education and will include reminders of the individualized goals set during the remote exercise intervention and consultation . The digital component will also offer a platform for patients to share their progress and seek further guidance during the scheduled in-person consultation. The use of digital AI feedback aligns with the trend of integrating technology into healthcare services, providing a convenient and accessible modality for supporting parents engaging in regular exercise.
  Arms: AI-PEF
Behavioral: Theory-based digital exercise — The theory-based digital exercise group will follow the same in-person clinic visits and walking program as AI-PEF but without AI-driven feedback
  Arms: Theory-based digital exercise
Behavioral: Active Control — Participants in the active control group will receive standard TBI care, including Garmin-based self-monitoring and routine clinic visits at baseline (T0), 3 months (T1), and 6 months (T2). These visits will include general health education and recommendations on daily physical activity. No personalized or digital exercise strategies will be provided. Participants completing the 6-month protocol will have the option to access the AI-PEF program after the study.
  Arms: Active control group

SUMMARY:
This study aims to develop and evaluate an AI-driven Personalized Exercise Feedback Program (AI-PEF) to enhance exercise adherence and health outcomes in mTBI patients.

Methods: AI-PEF integrates the transtheoretical model and self-determination theory with machine learning algorithms to provide real-time, personalized feedback. A phased randomized controlled trial will be conducted: Phase I evaluates feasibility and acceptability through Delphi methods with expert consensus and patient feedback; Phase II validates preliminary outcomes with 30 participants in a 2-arm randomized trial; and Phase III assesses the program's impact on adherence, sleep quality, depressive symptoms, and quality of life with 90 participants in a 3-arm randomized trial.

DETAILED DESCRIPTION:
The study will employ a stepwise, multi-phase design, combining a two- parallel-group pilot study and a three-arm randomized controlled trial (RCT) to evaluate the appropriateness, feasibility, acceptability, and effectiveness of the AI-PEF (Figure 5). Participants will be recruited from the neurosurgery clinics at Tri-Service General Hospital, Taipei. Recruitment will be facilitated through referrals by attending physicians and registered nurses, who will be briefed on the study protocol.

Study procedures

1. Phase I (Year 1): Development and Pilot Testing (Aim 1) Phase I will focus on developing and refining the AI-PEF through expert validation and pilot testing. This phase will use a sequential-parallel hybrid design to develop and evaluate the appropriateness of the AI-PEF to deliver personalized exercise empowerment. Stage 1, Delphi Process for AI-PEF Development: Ten experts from diverse fields will participate in two Delphi rounds to finalize the AI-PEF framework. This includes refining algorithms, educational materials, and preliminary validation of key components, such as personalization algorithms and behavior-change strategies. Stage 2, Small-Scale Pilot Study (Early Feedback): A single-arm pilot study with 5 patients will be conducted over four weeks to gather feedback on usability, engagement, and content clarity.
2. Phase II : Larger Pilot Study (Aim 2) Phase II will focus on evaluating the feasibility, acceptability, and preliminary effectiveness of the refined AI-PEF intervention. A two-parallel-group design will be employed, with 30 participants, 15 participants per group, randomly assigned in a 1:1 ratio to the AI-PEF group and Active control group. Over three months, AI-PEF participants will engage in personalized exercise guided by AI, while active control participants will follow standard exercise recommendations. Both qualitative and quantitative data will be collected. Assessments will occur at baseline (T0) and 3 months (T1), including fitness tracker data, questionnaires (motivation, sleep, symptoms), and semi-structured interviews. The primary outcome of interest will be adherence rates, while secondary outcomes will focus on motivation and various health metrics.
3. Phase III : Full- scale three-arm RCT (Aim 3) Phase III will assess the long-term impact of the AI- PEF on exercise adherence, motivation, and health outcomes through a 3-arm RCT randomly assigned to one of three groups: (1) the AI-PEF group, receiving a machine learning-powered personalized exercise program; (2) the Theory-based digital exercise group, engaging in structured digital exercise without machine learning- powered feedback; or (3) the Active control group, receiving general exercise recommendations as part of standard care in a 1:1:1 ratio. Over six months, participants will receive group-specific interventions, with assessments conducted at baseline (T0), 3 months (T1), and 6 months (T2). Primary outcomes, including exercise adherence, will be objectively measured via Garmin fitness trackers, while secondary outcomes, such as motivation, sleep quality, and symptom reduction, will be assessed through standardized questionnaires and qualitative interviews. These standardized questionnaires are being used in our current digital remote exercise trial in patients with mild TBI (NSTC 112-2314-B-016-007-MY2) and have performed well on physiological performance. Data will be collected and analyzed using both quantitative and qualitative methods to compare adherence, motivation, and health outcomes across the three groups, identifying the efficacy of AI-PEF relative to standard interventions. Procedures will adhere to the blinding and randomization protocols described in Intervention Fidelity, ensuring unbiased assignment and data collection processes. This proposed study protocol is closely aligned with those that have been successfully implemented in our previous digital exercise trial.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are patients aged over 18 with mild TBI (GCS 13-15)
* who can walk independently,
* reside in the Greater Taipei area,
* and possess sufficient Chinese or Taiwanese language proficiency to understand the trial
* complete self-administered questionnaires.

Exclusion Criteria:

* Exclusion criteria include individuals with severe medical conditions (e.g., respiratory failure, epilepsy, psychiatric disorders), musculoskeletal or neurological impairments
* hindering physical activity in the 6-minute walk test,
* cognitive impairments (MMSE < 24),
* frontal lobe injuries or penetrating injury causing significant psychological dysfunction.
* Patients regularly engaging in moderate-to-high-intensity aerobic exercise or participating in other studies will also be excluded to avoid bias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Adherence | T1-baseline
  Exercise adherence will be the primary outcome, defined as the percentage of participants completing at least five exercise sessions weekly over 12 weeks. Adherence will be objectively tracked using the Garmin Vivosmart 5, which monitors exercise duration and frequency. Range of adherence are 0- 100%, the higher percentage means the higher adherence.
Adherence | T2- 1 month later
  Exercise adherence will be the primary outcome, defined as the percentage of participants completing at least five exercise sessions weekly over 12 weeks. Adherence will be objectively tracked using the Garmin Vivosmart 5, which monitors exercise duration and frequency. Range of adherence are 0- 100%, the higher percentage means the higher adherence.
Adherence | T3- 2 month later
  Exercise adherence will be the primary outcome, defined as the percentage of participants completing at least five exercise sessions weekly over 12 weeks. Adherence will be objectively tracked using the Garmin Vivosmart 5, which monitors exercise duration and frequency. Range of adherence are 0- 100%, the higher percentage means the higher adherence.
Adherence | T4- 3 month later
  Exercise adherence will be the primary outcome, defined as the percentage of participants completing at least five exercise sessions weekly over 12 weeks. Adherence will be objectively tracked using the Garmin Vivosmart 5, which monitors exercise duration and frequency. Range of adherence are 0- 100%, the higher percentage means the higher adherence.
Adherence | T5- 6 month later
  Exercise adherence will be the primary outcome, defined as the percentage of participants completing at least five exercise sessions weekly over 12 weeks. Adherence will be objectively tracked using the Garmin Vivosmart 5, which monitors exercise duration and frequency. Range of adherence are 0- 100%, the higher percentage means the higher adherence.

SECONDARY OUTCOMES:
The Revised Sport Motivation Scale-II | T1- baseline
  The Revised Sport Motivation Scale-II (SMS-II), validated in Chinese, will measure six types of motivation, including amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. A total of 18 items with Likert scale 1-7, 5 domains: Intrinsic Regulation: 3, 9, 17, Integrated Regulation: 4, 11, 14, Identified Regulation: 6, 12, 18, Introjected Regulation: 1, 7, 16, External Regulation: 5, 8, 15, Non Regulation: 2, 10, 13. Each domain is record separately. The higher scores means the higher tendency of the domain. The range of the minimum and maximum values are 18-126.
The Revised Sport Motivation Scale-II | T2- 1 month later
  The Revised Sport Motivation Scale-II (SMS-II), validated in Chinese, will measure six types of motivation, including amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. A total of 18 items with Likert scale 1-7, 5 domains: Intrinsic Regulation: 3, 9, 17, Integrated Regulation: 4, 11, 14, Identified Regulation: 6, 12, 18, Introjected Regulation: 1, 7, 16, External Regulation: 5, 8, 15, Non Regulation: 2, 10, 13. Each domain is record separately. The higher scores means the higher tendency of the domain. The range of the minimum and maximum values are 18-126.
The Rivermead Post-Concussion Symptoms Questionnaire | T1 baseline
  The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) will assess physical, cognitive, and behavioral symptoms associated with TBI, validated for mild to moderate TBI cases. A total of 16 items, scored 0-4, ranged 0- 64, the higher scores mean the severity of the concussion symptoms.
The Beck Depression Inventory-II | T1 baseline
  The Beck Depression Inventory-II (BDI-II), with total scores categorized as follows: 0-13 (normal), 14-19 (mild depression), 20-28 (moderate depression), and 29-63 (severe depression), will evaluate depressive symptoms with established reliability (α = 0.94) and validity.
The Pittsburgh Sleep Quality Index | T1-baseline
  The Pittsburgh Sleep Quality Index (PSQI) will assess subjective sleep quality, using a validated Chinese version. Previous research has demonstrated good internal consistency reliability (0.82) and 14- to 21-day test-retest reliability (0.85) of the PSQI Chinese version in Taiwan's populations. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties.
The Godin-Shephard Leisure Time Physical Activity Questionnaire | T1 -baseline
  The Godin-Shephard Leisure Time Physical Activity Questionnaire (GLTPA) will measure weekly physical activity intensity, classified into light, moderate, and vigorous levels. The Chinese version of the GLTPA has shown good validity and is significantly correlated with mental health outcomes. By classifying physical activity intensity lasting for more than 15 minutes in the past week into strenuous activities, moderate strenuous activities, and light activities, and then multiplying by corresponding coefficients 9, 5, and 3 respectively for quantification, the sum of these scores is Godin's leisure time physical Total activity score, with higher scores indicating greater physical activity. The level of physical activity can be divided into three levels according to the total Godin leisure time physical activity score. A total score of 24 or above is considered active, a score between 14 and 23 is moderately active, and a score below 14 is consider Insufficiently active.
The World Health Organization Quality of Life Scale-brief | T1 - baseline
  The World Health Organization Quality of Life Scale-brief (WHOQOL-BREF), validated in Chinese, with good internal consistency (α = 0.70-0.77), overall reliability (α = 0.91), and test-retest reliability (0.76-0.80), will assess the quality of life across four domains: physical, psychological, social, and environmental well-being. This scale covers subjective life feelings in four major categories: physical health, psychological, social relations, and environment. It has 24 questions in total. There are also 2 questions measuring the overall quality of life and general health at the general level. (general health), in addition, the Taiwan version adds 2 local questions, namely diet (whether you can eat the food you want) and face issues (whether you are respected), a total of 28 questions, and the scores for each category are introduced. Between 4 and 20, the higher the score, the better the quality of life.
Advanced sleep pattern | T1- baseline
  Garmin Vivosmart 5. This wearable device will track heart rate, exercise intensity, and sleep patterns. HR will be track every second. Advanced sleep tracking in compatible Garmin devices takes into account multiple factors to help understanding of sleep. In addition to the basics, such as when participants fell asleep and when they woke up, researchers can see times when they were awake and how much time they spent in key sleep stages (light, deep, REM), and the data will be calculated by heart rate to increase its validity.
Mini-Mental State Examination | T1- baseline
  Cognitive function will be assessed pre-enrollment using the MMSE, with validated age- and education-adjusted thresholds. The MMSE has demonstrated good reliability and validity and is a strong predictor of disability levels in patients with traumatic brain injury. Participants with an MMSE score below 24 will be excluded from the study to ensure appropriate cognitive capacity for participation. The score range is 0-30 points, with the international standard cut-off value of 24 points, 18-24 points as mild dementia, 16-17 points as moderate dementia, and ≦15 points as severe dementia.
6-Minute Walk Test | T1-baseline
  Cardiorespiratory fitness will be evaluated using the 6MWT, measuring the distance walked in six minutes as a reliable indicator of endurance. The higher distance means better cardiorespiratory fitness.
The mHealth App usability questionnaire | T1-baseline
  The Mobile App Usability Questionnaire (MAUQ) assesses usability across three dimensions: usability and satisfaction, system information arrangement, and system efficiency. A Chinese version of the questionnaire was developed in 2022, with an internal consistency reliability (Cronbach's α) of 0.988 and an internal consistency range of 0.845-0.931. The test-retest reliability ranges from 0.828 to 0.918. A total of 21 items, Likert scale scores ranged from 1 (strongly agree) to 7 (strongly disagree), indicating the lower scores the better usability.
Montreal Cognitive Assessment | T1-baseline
  The Montreal Cognitive Assessment (MoCA) is a sensitive tool for the early screening of mild cognitive impairment, particularly useful for detecting deficits in executive function, attention, short-term memory, language fluency, abstract thinking, and visuospatial abilities. The total score of the scale is 30 points, with a score of less than 26 considered indicative of possible mild cognitive impairment. The score can be adjusted (+1 point) based on educational level. The Chinese version of MoCA has been proven to have good reliability and validity (Cronbach's α = 0.83) and is particularly suitable for research populations in Asian regions.
Near-Infrared Brain Blood Flow Imaging | T1 - baseline
  In this study, the Biolight MediTECH® near-infrared brain blood flow imaging sensor (hemoencephalography; HEG) was used to measure blood flow in the prefrontal cortex. The Biolight near-infrared spectroscopy device is an HEG sensor designed by MediTECH®, based on NIR technology to observe the optical properties of cells and tissues at the reflection level. This enables monitoring of changes in oxyhemoglobin and deoxyhemoglobin concentrations. By measuring light absorption at different wavelengths, the system can continuously track changes during tissue oxidation processes, thereby measuring cerebral blood flow conditions. The percentage of the NIR brain blood flow ranged 0- 100%, the higher percentage means the higher prefrontal brain blood flow.
cardiac metabolic performance benchmark | T1- baseline
  Preliminary findings from this study applied the cardiac metabolic performance benchmark (CMPB3) to compare the effectiveness of increasing cerebral blood circulation at different intensities (CMPB3 ≤ 35, 40, 45, 50). Results indicated that CMPB3 levels above 40 effectively increased cerebral blood circulation, with improvements observed not only during exercise but also during the post-exercise rest period, where cerebral blood flow remained higher than the baseline level. The lower intensity means the lower exercise intensity and the higher ability to perform aerobic walking exercise. The benchmark will be calculated by the Heart rate measured by Garmin fitness bracelet.
Semi-Structured Interviews | T1- baseline
  This study will adopt semi-structured interviews to gain an in-depth understanding of participants' experiences and perceptions of the walking program, as well as to complement and interpret quantitative data.
  It is a qualitative data, not a quantitative data.
  The interview content covers three major themes:
  1. Benefits of the walking program;
  2. Experiences and challenges of the walking program;
  3. The impact of the walking program on quality of life, sleep quality, concussion symptoms, psychological resilience, depression, exercise motivation, exercise self-efficacy, and physical activity.
The Revised Sport Motivation Scale-II | T3- 2 month later
  The Revised Sport Motivation Scale-II (SMS-II), validated in Chinese, will measure six types of motivation, including amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. A total of 18 items with Likert scale 1-7, 5 domains: Intrinsic Regulation: 3, 9, 17, Integrated Regulation: 4, 11, 14, Identified Regulation: 6, 12, 18, Introjected Regulation: 1, 7, 16, External Regulation: 5, 8, 15, Non Regulation: 2, 10, 13. Each domain is record separately. The higher scores means the higher tendency of the domain. The range of the minimum and maximum values are 18-126.
The Revised Sport Motivation Scale-II | T4- 3 month later
  The Revised Sport Motivation Scale-II (SMS-II), validated in Chinese, will measure six types of motivation, including amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. A total of 18 items with Likert scale 1-7, 5 domains: Intrinsic Regulation: 3, 9, 17, Integrated Regulation: 4, 11, 14, Identified Regulation: 6, 12, 18, Introjected Regulation: 1, 7, 16, External Regulation: 5, 8, 15, Non Regulation: 2, 10, 13. Each domain is record separately. The higher scores means the higher tendency of the domain. The range of the minimum and maximum values are 18-126.
The Revised Sport Motivation Scale-II | T5- 6 month later
  The Revised Sport Motivation Scale-II (SMS-II), validated in Chinese, will measure six types of motivation, including amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic motivation. A total of 18 items with Likert scale 1-7, 5 domains: Intrinsic Regulation: 3, 9, 17, Integrated Regulation: 4, 11, 14, Identified Regulation: 6, 12, 18, Introjected Regulation: 1, 7, 16, External Regulation: 5, 8, 15, Non Regulation: 2, 10, 13. Each domain is record separately. The higher scores means the higher tendency of the domain. The range of the minimum and maximum values are 18-126.
The Rivermead Post-Concussion Symptoms Questionnaire | T2 1 month later
  The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) will assess physical, cognitive, and behavioral symptoms associated with TBI, validated for mild to moderate TBI cases. A total of 16 items, scored 0-4, ranged 0- 64, the higher scores mean the severity of the concussion symptoms.
The Rivermead Post-Concussion Symptoms Questionnaire | T3 2 month later
  The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) will assess physical, cognitive, and behavioral symptoms associated with TBI, validated for mild to moderate TBI cases. A total of 16 items, scored 0-4, ranged 0- 64, the higher scores mean the severity of the concussion symptoms.
The Rivermead Post-Concussion Symptoms Questionnaire | T4 3 month later
  The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) will assess physical, cognitive, and behavioral symptoms associated with TBI, validated for mild to moderate TBI cases. A total of 16 items, scored 0-4, ranged 0- 64, the higher scores mean the severity of the concussion symptoms.
The Rivermead Post-Concussion Symptoms Questionnaire | T5 6 month
  The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) will assess physical, cognitive, and behavioral symptoms associated with TBI, validated for mild to moderate TBI cases. A total of 16 items, scored 0-4, ranged 0- 64, the higher scores mean the severity of the concussion symptoms.
The Beck Depression Inventory-II | T2 1 month later
  The Beck Depression Inventory-II (BDI-II), with total scores categorized as follows: 0-13 (normal), 14-19 (mild depression), 20-28 (moderate depression), and 29-63 (severe depression), will evaluate depressive symptoms with established reliability (α = 0.94) and validity.
The Beck Depression Inventory-II | T3 2 month later
  The Beck Depression Inventory-II (BDI-II), with total scores categorized as follows: 0-13 (normal), 14-19 (mild depression), 20-28 (moderate depression), and 29-63 (severe depression), will evaluate depressive symptoms with established reliability (α = 0.94) and validity.
The Beck Depression Inventory-II | T4-3 month later
  The Beck Depression Inventory-II (BDI-II), with total scores categorized as follows: 0-13 (normal), 14-19 (mild depression), 20-28 (moderate depression), and 29-63 (severe depression), will evaluate depressive symptoms with established reliability (α = 0.94) and validity.
The Beck Depression Inventory-II | T5- 6 month later
  The Beck Depression Inventory-II (BDI-II), with total scores categorized as follows: 0-13 (normal), 14-19 (mild depression), 20-28 (moderate depression), and 29-63 (severe depression), will evaluate depressive symptoms with established reliability (α = 0.94) and validity.
The Pittsburgh Sleep Quality Index | T2- 1 month later
  The Pittsburgh Sleep Quality Index (PSQI) will assess subjective sleep quality, using a validated Chinese version [68]. Previous research has demonstrated good internal consistency reliability (0.82) and 14- to 21-day test-retest reliability (0.85) of the PSQI Chinese version in Taiwan's populations. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
The Pittsburgh Sleep Quality Index | T3-2 month later
  The Pittsburgh Sleep Quality Index (PSQI) will assess subjective sleep quality, using a validated Chinese version [68]. Previous research has demonstrated good internal consistency reliability (0.82) and 14- to 21-day test-retest reliability (0.85) of the PSQI Chinese version in Taiwan's populations. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
The Pittsburgh Sleep Quality Index | T4-3 month later
  The Pittsburgh Sleep Quality Index (PSQI) will assess subjective sleep quality, using a validated Chinese version [68]. Previous research has demonstrated good internal consistency reliability (0.82) and 14- to 21-day test-retest reliability (0.85) of the PSQI Chinese version in Taiwan's populations. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
The Pittsburgh Sleep Quality Index | T5-6 month later
  The Pittsburgh Sleep Quality Index (PSQI) will assess subjective sleep quality, using a validated Chinese version [68]. Previous research has demonstrated good internal consistency reliability (0.82) and 14- to 21-day test-retest reliability (0.85) of the PSQI Chinese version in Taiwan's populations. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
The Godin-Shephard Leisure Time Physical Activity Questionnaire | T2 -1 month later
  The Godin-Shephard Leisure Time Physical Activity Questionnaire (GLTPA) will measure weekly physical activity intensity, classified into light, moderate, and vigorous levels. The Chinese version of the GLTPA has shown good validity and is significantly correlated with mental health outcomes. By classifying physical activity intensity lasting for more than 15 minutes in the past week into strenuous activities, moderate strenuous activities, and light activities, and then multiplying by corresponding coefficients 9, 5, and 3 respectively for quantification, the sum of these scores is Godin's leisure time physical Total activity score, with higher scores indicating greater physical activity. The level of physical activity can be divided into three levels according to the total Godin leisure time physical activity score. A total score of 24 or above is considered active, a score between 14 and 23 is moderately active, and a score below 14 is consider Insufficiently active .
The Godin-Shephard Leisure Time Physical Activity Questionnaire | T3 -2 month later
  The Godin-Shephard Leisure Time Physical Activity Questionnaire (GLTPA) will measure weekly physical activity intensity, classified into light, moderate, and vigorous levels. The Chinese version of the GLTPA has shown good validity and is significantly correlated with mental health outcomes. By classifying physical activity intensity lasting for more than 15 minutes in the past week into strenuous activities, moderate strenuous activities, and light activities, and then multiplying by corresponding coefficients 9, 5, and 3 respectively for quantification, the sum of these scores is Godin's leisure time physical Total activity score, with higher scores indicating greater physical activity. The level of physical activity can be divided into three levels according to the total Godin leisure time physical activity score. A total score of 24 or above is considered active, a score between 14 and 23 is moderately active, and a score below 14 is consider Insufficiently active.
The Godin-Shephard Leisure Time Physical Activity Questionnaire | T4-3 month later
  The Godin-Shephard Leisure Time Physical Activity Questionnaire (GLTPA) will measure weekly physical activity intensity, classified into light, moderate, and vigorous levels. The Chinese version of the GLTPA has shown good validity and is significantly correlated with mental health outcomes. By classifying physical activity intensity lasting for more than 15 minutes in the past week into strenuous activities, moderate strenuous activities, and light activities, and then multiplying by corresponding coefficients 9, 5, and 3 respectively for quantification, the sum of these scores is Godin's leisure time physical Total activity score, with higher scores indicating greater physical activity. The level of physical activity can be divided into three levels according to the total Godin leisure time physical activity score. A total score of 24 or above is considered active, a score between 14 and 23 is moderately active, and a score below 14 is consider Insufficiently active.
The Godin-Shephard Leisure Time Physical Activity Questionnaire | T5-6 month later
  The Godin-Shephard Leisure Time Physical Activity Questionnaire (GLTPA) will measure weekly physical activity intensity, classified into light, moderate, and vigorous levels. The Chinese version of the GLTPA has shown good validity and is significantly correlated with mental health outcomes. By classifying physical activity intensity lasting for more than 15 minutes in the past week into strenuous activities, moderate strenuous activities, and light activities, and then multiplying by corresponding coefficients 9, 5, and 3 respectively for quantification, the sum of these scores is Godin's leisure time physical Total activity score, with higher scores indicating greater physical activity. The level of physical activity can be divided into three levels according to the total Godin leisure time physical activity score. A total score of 24 or above is considered active, a score between 14 and 23 is moderately active, and a score below 14 is consider Insufficiently active.
The World Health Organization Quality of Life Scale-brief | T2 - 1 month later
  The World Health Organization Quality of Life Scale-brief (WHOQOL-BREF), validated in Chinese, with good internal consistency (α = 0.70-0.77), overall reliability (α = 0.91), and test-retest reliability (0.76-0.80), will assess the quality of life across four domains: physical, psychological, social, and environmental well-being. This scale covers subjective life feelings in four major categories: physical health, psychological, social relations, and environment. It has 24 questions in total. There are also 2 questions measuring the overall quality of life and general health at the general level. (general health), in addition, the Taiwan version adds 2 local questions, namely diet (whether you can eat the food you want) and face issues (whether you are respected), a total of 28 questions, and the scores for each category are introduced. Between 4 and 20, the higher the score, the better the quality of life.
The World Health Organization Quality of Life Scale-brief | T3 - 2 month later
  The World Health Organization Quality of Life Scale-brief (WHOQOL-BREF), validated in Chinese, with good internal consistency (α = 0.70-0.77), overall reliability (α = 0.91), and test-retest reliability (0.76-0.80), will assess the quality of life across four domains: physical, psychological, social, and environmental well-being. This scale covers subjective life feelings in four major categories: physical health, psychological, social relations, and environment. It has 24 questions in total. There are also 2 questions measuring the overall quality of life and general health at the general level. (general health), in addition, the Taiwan version adds 2 local questions, namely diet (whether you can eat the food you want) and face issues (whether you are respected), a total of 28 questions, and the scores for each category are introduced. Between 4 and 20, the higher the score, the better the quality of life.
The World Health Organization Quality of Life Scale-brief | T4 - 3 month later
  The World Health Organization Quality of Life Scale-brief (WHOQOL-BREF), validated in Chinese, with good internal consistency (α = 0.70-0.77), overall reliability (α = 0.91), and test-retest reliability (0.76-0.80), will assess the quality of life across four domains: physical, psychological, social, and environmental well-being. This scale covers subjective life feelings in four major categories: physical health, psychological, social relations, and environment. It has 24 questions in total. There are also 2 questions measuring the overall quality of life and general health at the general level. (general health), in addition, the Taiwan version adds 2 local questions, namely diet (whether you can eat the food you want) and face issues (whether you are respected), a total of 28 questions, and the scores for each category are introduced. Between 4 and 20, the higher the score, the better the quality of life.
The World Health Organization Quality of Life Scale-brief | T5- 6 month later
  The World Health Organization Quality of Life Scale-brief (WHOQOL-BREF), validated in Chinese, with good internal consistency (α = 0.70-0.77), overall reliability (α = 0.91), and test-retest reliability (0.76-0.80), will assess the quality of life across four domains: physical, psychological, social, and environmental well-being. This scale covers subjective life feelings in four major categories: physical health, psychological, social relations, and environment. It has 24 questions in total. There are also 2 questions measuring the overall quality of life and general health at the general level. (general health), in addition, the Taiwan version adds 2 local questions, namely diet (whether you can eat the food you want) and face issues (whether you are respected), a total of 28 questions, and the scores for each category are introduced. Between 4 and 20, the higher the score, the better the quality of life.
Mini-Mental State Examination | T2-1 month later
  Cognitive function will be assessed pre-enrollment using the MMSE, with validated age- and education-adjusted thresholds [75]. The MMSE has demonstrated good reliability and validity and is a strong predictor of disability levels in patients with traumatic brain injury [76]. Participants with an MMSE score below 24 will be excluded from the study to ensure appropriate cognitive capacity for participation. The score range is 0-30 points, with the international standard cut-off value of 24 points, 18-24 points as mild dementia, 16-17 points as moderate dementia, and ≦15 points as severe dementia.
Mini-Mental State Examination | T3-2 month later
  Cognitive function will be assessed pre-enrollment using the MMSE, with validated age- and education-adjusted thresholds [75]. The MMSE has demonstrated good reliability and validity and is a strong predictor of disability levels in patients with traumatic brain injury [76]. Participants with an MMSE score below 24 will be excluded from the study to ensure appropriate cognitive capacity for participation. The score range is 0-30 points, with the international standard cut-off value of 24 points, 18-24 points as mild dementia, 16-17 points as moderate dementia, and ≦15 points as severe dementia.
Mini-Mental State Examination | T4-3 month later
  Cognitive function will be assessed pre-enrollment using the MMSE, with validated age- and education-adjusted thresholds. The MMSE has demonstrated good reliability and validity and is a strong predictor of disability levels in patients with traumatic brain injury. Participants with an MMSE score below 24 will be excluded from the study to ensure appropriate cognitive capacity for participation. The score range is 0-30 points, with the international standard cut-off value of 24 points, 18-24 points as mild dementia, 16-17 points as moderate dementia, and ≦15 points as severe dementia.
Mini-Mental State Examination | T5- 6 month later
  Cognitive function will be assessed pre-enrollment using the MMSE, with validated age- and education-adjusted thresholds. The MMSE has demonstrated good reliability and validity and is a strong predictor of disability levels in patients with traumatic brain injury. Participants with an MMSE score below 24 will be excluded from the study to ensure appropriate cognitive capacity for participation. The score range is 0-30 points, with the international standard cut-off value of 24 points, 18-24 points as mild dementia, 16-17 points as moderate dementia, and ≦15 points as severe dementia.
6-Minute Walk Test | T2-1 month later
  Cardiorespiratory fitness will be evaluated using the 6MWT, measuring the distance walked in six minutes as a reliable indicator of endurance. The higher distance means better cardiorespiratory fitness.
6-Minute Walk Test | T3- 2 month later
  Cardiorespiratory fitness will be evaluated using the 6MWT, measuring the distance walked in six minutes as a reliable indicator of endurance. The higher distance means better cardiorespiratory fitness.
6-Minute Walk Test | T4-3 month later
  Cardiorespiratory fitness will be evaluated using the 6MWT, measuring the distance walked in six minutes as a reliable indicator of endurance. The higher distance means better cardiorespiratory fitness.
6-Minute Walk Test | T1-baseline
  Cardiorespiratory fitness will be evaluated using the 6-Minute Walk Test (6MWT), measuring the distance walked in six minutes as a reliable indicator of endurance. The higher distance means better cardiorespiratory fitness.
The mHealth App usability questionnaire | T2- 1 month
  The Mobile App Usability Questionnaire (MAUQ) assesses usability across three dimensions: usability and satisfaction, system information arrangement, and system efficiency. A Chinese version of the questionnaire was developed in 2022, with an internal consistency reliability (Cronbach's α) of 0.988 and an internal consistency range of 0.845-0.931. The test-retest reliability ranges from 0.828 to 0.918. A total of 21 items, Likert scale scores ranged from 1 (strongly agree) to 7 (strongly disagree), indicating the lower scores the better usability.
The mHealth App usability questionnaire | T3-2 month later
  The Mobile App Usability Questionnaire (MAUQ) assesses usability across three dimensions: usability and satisfaction, system information arrangement, and system efficiency. A Chinese version of the questionnaire was developed in 2022, with an internal consistency reliability (Cronbach's α) of 0.988 and an internal consistency range of 0.845-0.931. The test-retest reliability ranges from 0.828 to 0.918. A total of 21 items, Likert scale scores ranged from 1 (strongly agree) to 7 (strongly disagree), indicating the lower scores the better usability.
The mHealth App usability questionnaire | T4-3 month later
  The Mobile App Usability Questionnaire (MAUQ) assesses usability across three dimensions: usability and satisfaction, system information arrangement, and system efficiency. A Chinese version of the questionnaire was developed in 2022, with an internal consistency reliability (Cronbach's α) of 0.988 and an internal consistency range of 0.845-0.931. The test-retest reliability ranges from 0.828 to 0.918. A total of 21 items, Likert scale scores ranged from 1 (strongly agree) to 7 (strongly disagree), indicating the lower scores the better usability.
The mHealth App usability questionnaire | T5-6 month later
  The Mobile App Usability Questionnaire (MAUQ) assesses usability across three dimensions: usability and satisfaction, system information arrangement, and system efficiency. A Chinese version of the questionnaire was developed in 2022, with an internal consistency reliability (Cronbach's α) of 0.988 and an internal consistency range of 0.845-0.931. The test-retest reliability ranges from 0.828 to 0.918. A total of 21 items, Likert scale scores ranged from 1 (strongly agree) to 7 (strongly disagree), indicating the lower scores the better usability.
Montreal Cognitive Assessment | T2-1 month later
  The Montreal Cognitive Assessment (MoCA) is a sensitive tool for the early screening of mild cognitive impairment, particularly useful for detecting deficits in executive function, attention, short-term memory, language fluency, abstract thinking, and visuospatial abilities. The total score of the scale is 30 points, with a score of less than 26 considered indicative of possible mild cognitive impairment. The score can be adjusted (+1 point) based on educational level. The Chinese version of MoCA has been proven to have good reliability and validity (Cronbach's α = 0.83) and is particularly suitable for research populations in Asian regions.
Montreal Cognitive Assessment | T3-2 month later
  The Montreal Cognitive Assessment (MoCA) is a sensitive tool for the early screening of mild cognitive impairment, particularly useful for detecting deficits in executive function, attention, short-term memory, language fluency, abstract thinking, and visuospatial abilities. The total score of the scale is 30 points, with a score of less than 26 considered indicative of possible mild cognitive impairment. The score can be adjusted (+1 point) based on educational level. The Chinese version of MoCA has been proven to have good reliability and validity (Cronbach's α = 0.83) and is particularly suitable for research populations in Asian regions.
Montreal Cognitive Assessment | T4-3 month later
  The Montreal Cognitive Assessment (MoCA) is a sensitive tool for the early screening of mild cognitive impairment, particularly useful for detecting deficits in executive function, attention, short-term memory, language fluency, abstract thinking, and visuospatial abilities. The total score of the scale is 30 points, with a score of less than 26 considered indicative of possible mild cognitive impairment. The score can be adjusted (+1 point) based on educational level. The Chinese version of MoCA has been proven to have good reliability and validity (Cronbach's α = 0.83) and is particularly suitable for research populations in Asian regions.
Montreal Cognitive Assessment | T5-6 month later
  The Montreal Cognitive Assessment (MoCA) is a sensitive tool for the early screening of mild cognitive impairment, particularly useful for detecting deficits in executive function, attention, short-term memory, language fluency, abstract thinking, and visuospatial abilities. The total score of the scale is 30 points, with a score of less than 26 considered indicative of possible mild cognitive impairment. The score can be adjusted (+1 point) based on educational level. The Chinese version of MoCA has been proven to have good reliability and validity (Cronbach's α = 0.83) and is particularly suitable for research populations in Asian regions.
Near-Infrared Brain Blood Flow Imaging | T2- 1 month later
  In this study, the Biolight MediTECH® near-infrared brain blood flow imaging sensor (hemoencephalography; HEG) was used to measure blood flow in the prefrontal cortex. The Biolight near-infrared spectroscopy device is an HEG sensor designed by MediTECH®, based on NIR technology to observe the optical properties of cells and tissues at the reflection level. This enables monitoring of changes in oxyhemoglobin and deoxyhemoglobin concentrations. By measuring light absorption at different wavelengths, the system can continuously track changes during tissue oxidation processes, thereby measuring cerebral blood flow conditions. The percentage of the NIR brain blood flow ranged 0- 100%, the higher percentage means the higher prefrontal brain blood flow.
Near-Infrared Brain Blood Flow Imaging | T3-2 month later
  In this study, the Biolight MediTECH® near-infrared brain blood flow imaging sensor (hemoencephalography; HEG) was used to measure blood flow in the prefrontal cortex. The Biolight near-infrared spectroscopy device is an HEG sensor designed by MediTECH®, based on NIR technology to observe the optical properties of cells and tissues at the reflection level. This enables monitoring of changes in oxyhemoglobin and deoxyhemoglobin concentrations. By measuring light absorption at different wavelengths, the system can continuously track changes during tissue oxidation processes, thereby measuring cerebral blood flow conditions. The percentage of the NIR brain blood flow ranged 0- 100%, the higher percentage means the higher prefrontal brain blood flow.
Near-Infrared Brain Blood Flow Imaging | T4- 3 month later
  In this study, the Biolight MediTECH® near-infrared brain blood flow imaging sensor (hemoencephalography; HEG) was used to measure blood flow in the prefrontal cortex. The Biolight near-infrared spectroscopy device is an HEG sensor designed by MediTECH®, based on NIR technology to observe the optical properties of cells and tissues at the reflection level. This enables monitoring of changes in oxyhemoglobin and deoxyhemoglobin concentrations. By measuring light absorption at different wavelengths, the system can continuously track changes during tissue oxidation processes, thereby measuring cerebral blood flow conditions. The percentage of the NIR brain blood flow ranged 0- 100%, the higher percentage means the higher prefrontal brain blood flow.
Near-Infrared Brain Blood Flow Imaging | T5- 6 month later
  In this study, the Biolight MediTECH® near-infrared brain blood flow imaging sensor (hemoencephalography; HEG) was used to measure blood flow in the prefrontal cortex. The Biolight near-infrared spectroscopy device is an HEG sensor designed by MediTECH®, based on NIR technology to observe the optical properties of cells and tissues at the reflection level. This enables monitoring of changes in oxyhemoglobin and deoxyhemoglobin concentrations. By measuring light absorption at different wavelengths, the system can continuously track changes during tissue oxidation processes, thereby measuring cerebral blood flow conditions. The percentage of the NIR brain blood flow ranged 0- 100%, the higher percentage means the higher prefrontal brain blood flow.
cardiac metabolic performance benchmark | T2- 1 month later
  Preliminary findings from this study applied the cardiac metabolic performance benchmark (CMPB3) to compare the effectiveness of increasing cerebral blood circulation at different intensities (CMPB3 ≤ 35, 40, 45, 50). Results indicated that CMPB3 levels above 40 effectively increased cerebral blood circulation, with improvements observed not only during exercise but also during the post-exercise rest period, where cerebral blood flow remained higher than the baseline level. The lower intensity means the lower exercise intensity and the higher ability to perform aerobic walking exercise.
cardiac metabolic performance benchmark | T3-2 month later
  Preliminary findings from this study applied the cardiac metabolic performance benchmark (CMPB3) to compare the effectiveness of increasing cerebral blood circulation at different intensities (CMPB3 ≤ 35, 40, 45, 50). Results indicated that CMPB3 levels above 40 effectively increased cerebral blood circulation, with improvements observed not only during exercise but also during the post-exercise rest period, where cerebral blood flow remained higher than the baseline level. The lower intensity means the lower exercise intensity and the higher ability to perform aerobic walking exercise.
cardiac metabolic performance benchmark | T4- 3 month later
  Preliminary findings from this study applied the cardiac metabolic performance benchmark (CMPB3) to compare the effectiveness of increasing cerebral blood circulation at different intensities (CMPB3 ≤ 35, 40, 45, 50). Results indicated that CMPB3 levels above 40 effectively increased cerebral blood circulation, with improvements observed not only during exercise but also during the post-exercise rest period, where cerebral blood flow remained higher than the baseline level. The lower intensity means the lower exercise intensity and the higher ability to perform aerobic walking exercise.
cardiac metabolic performance benchmark | T5- 6 month later
  Preliminary findings from this study applied the cardiac metabolic performance benchmark (CMPB3) to compare the effectiveness of increasing cerebral blood circulation at different intensities (CMPB3 ≤ 35, 40, 45, 50). Results indicated that CMPB3 levels above 40 effectively increased cerebral blood circulation, with improvements observed not only during exercise but also during the post-exercise rest period, where cerebral blood flow remained higher than the baseline level. The lower intensity means the lower exercise intensity and the higher ability to perform aerobic walking exercise.
Semi-Structured Interviews | T2- 1 month later
  This study will adopt semi-structured interviews to gain an in-depth understanding of participants' experiences and perceptions of the walking program, as well as to complement and interpret quantitative data.
  It is a qualitative data, not a quantitative data.
  The interview content covers three major themes:
  1. Benefits of the walking program;
  2. Experiences and challenges of the walking program;
  3. The impact of the walking program on quality of life, sleep quality, concussion symptoms, psychological resilience, depression, exercise motivation, exercise self-efficacy, and physical activity.
Semi-Structured Interviews | T3- 2 month later
  This study will adopt semi-structured interviews to gain an in-depth understanding of participants' experiences and perceptions of the walking program, as well as to complement and interpret quantitative data.
  It is a qualitative data, not a quantitative data.
  The interview content covers three major themes:
  1. Benefits of the walking program;
  2. Experiences and challenges of the walking program;
  3. The impact of the walking program on quality of life, sleep quality, concussion symptoms, psychological resilience, depression, exercise motivation, exercise self-efficacy, and physical activity.
Semi-Structured Interviews | T4-3 month later
  This study will adopt semi-structured interviews to gain an in-depth understanding of participants' experiences and perceptions of the walking program, as well as to complement and interpret quantitative data.
  It is a qualitative data, not a quantitative data.
  The interview content covers three major themes:
  1. Benefits of the walking program;
  2. Experiences and challenges of the walking program;
  3. The impact of the walking program on quality of life, sleep quality, concussion symptoms, psychological resilience, depression, exercise motivation, exercise self-efficacy, and physical activity.
Semi-Structured Interviews | T5- 6 month later
  This study will adopt semi-structured interviews to gain an in-depth understanding of participants' experiences and perceptions of the walking program, as well as to complement and interpret quantitative data.
  It is a qualitative data, not a quantitative data.
  The interview content covers three major themes:
  1. Benefits of the walking program;
  2. Experiences and challenges of the walking program;
  3. The impact of the walking program on quality of life, sleep quality, concussion symptoms, psychological resilience, depression, exercise motivation, exercise self-efficacy, and physical activity.
Physiological Monitoring Tools | T2- 1 month later
  Garmin Vivosmart 5. This wearable device will track heart rate, exercise intensity, and sleep patterns. Data will be integrated with the Garmin Connect app for real-time monitoring and feedback. Through our preliminary study conducted by the research team in 2020 showed a high correlation (r = 0.91) between the heart rate measurements of the Garmin Vivosmart and the Zephyr BioHarness, validating its accuracy for home-based heart rate monitoring. Participants will wear the device at home to facilitate real-time tracking of exercise intensity and physiological responses during the intervention. HR will be track every second. Advanced sleep tracking in compatible Garmin devices takes into account multiple factors to help understanding of sleep. In addition to the basics, such as when participants fell asleep and when they woke up, researchers can see times when they were awake and how much time they spent in key sleep stages (light, deep, REM).
Physiological Monitoring Tools | T3-2 month later
  Garmin Vivosmart 5. This wearable device will track heart rate, exercise intensity, and sleep patterns. Data will be integrated with the Garmin Connect app for real-time monitoring and feedback. Through our preliminary study conducted by the research team in 2020 showed a high correlation (r = 0.91) between the heart rate measurements of the Garmin Vivosmart and the Zephyr BioHarness, validating its accuracy for home-based heart rate monitoring. Participants will wear the device at home to facilitate real-time tracking of exercise intensity and physiological responses during the intervention. HR will be track every second. Advanced sleep tracking in compatible Garmin devices takes into account multiple factors to help understanding of sleep. In addition to the basics, such as when participants fell asleep and when they woke up, researchers can see times when they were awake and how much time they spent in key sleep stages (light, deep, REM).
Physiological Monitoring Tools | T4-3 month later
  Garmin Vivosmart 5. This wearable device will track heart rate, exercise intensity, and sleep patterns. Data will be integrated with the Garmin Connect app for real-time monitoring and feedback. Through our preliminary study conducted by the research team in 2020 showed a high correlation (r = 0.91) between the heart rate measurements of the Garmin Vivosmart and the Zephyr BioHarness, validating its accuracy for home-based heart rate monitoring. Participants will wear the device at home to facilitate real-time tracking of exercise intensity and physiological responses during the intervention. HR will be track every second. Advanced sleep tracking in compatible Garmin devices takes into account multiple factors to help understanding of sleep. In addition to the basics, such as when participants fell asleep and when they woke up, researchers can see times when they were awake and how much time they spent in key sleep stages (light, deep, REM).
Physiological Monitoring Tools | T5- 6 month later
  Garmin Vivosmart 5. This wearable device will track heart rate, exercise intensity, and sleep patterns. Data will be integrated with the Garmin Connect app for real-time monitoring and feedback. Through our preliminary study conducted by the research team in 2020 showed a high correlation (r = 0.91) between the heart rate measurements of the Garmin Vivosmart and the Zephyr BioHarness, validating its accuracy for home-based heart rate monitoring. Participants will wear the device at home to facilitate real-time tracking of exercise intensity and physiological responses during the intervention. HR will be track every second. Advanced sleep tracking in compatible Garmin devices takes into account multiple factors to help understanding of sleep. In addition to the basics, such as when participants fell asleep and when they woke up, researchers can see times when they were awake and how much time they spent in key sleep stages (light, deep, REM).

IPD SHARING:
Plan to Share IPD: No